CLINICAL TRIAL: NCT07081828
Title: The Asensus Paediatric Registry of Robotic-Assisted Endoscopic Procedures in Urology, Gynaecology, and General Surgery
Brief Title: The Asensus Paediatric Robotic Registry
Acronym: miniTRUST
Status: Recruiting | Type: Observational
Sponsor: Asensus Surgical (Industry)
Collaborators: RQM+ (Industry)
Responsible Party: Sponsor
Other Study IDs: miniTRUST
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Surgery; Surgery in Early Childhood
Keywords: Robotic; Laparoscopic; Senhance
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Surgery — Patients who undergo surgery utilising the Senhance Surgical System.

SUMMARY:
An open-label, observational, paediatric registry trial in which participating centers enroll subjects who had or will have a laparoscopically-assisted surgery using the Senhance Surgical System.

DETAILED DESCRIPTION:
This is a prospective and retrospective, multi-center, observational registry study evaluating the use of the Senhance Surgical System in paediatric patients undergoing laparoscopically-assisted surgery. The trial is open-label and designed to collect both historical and prospective data from participating centers. Paediatric subjects who have undergone or will undergo procedures with the Senhance Surgical System will be enrolled. The primary purpose for this study is to assess safety outcomes. Secondary endpoints include length of hospital stay, procedural information, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years of age
* Body weight > 10 kg
* Indication for a potential robot-assisted operation
* Expected survival of > 3 months

Exclusion Criteria:

* Subjects requiring surgery on the heart or greater vessels.
* Subjects for whom a laparoscopic approach and endoscopic approach in the thoracic area is not appropriate.
* Anaesthetic contraindications, children with pacemakers or other implants for which electrosurgery must be avoided, children with cancer, parents who prefer to proceed with classical or manual laparoscopic surgery.
* Subjects pregnant over the second trimester of pregnancy.
* Parents or children with insufficient understanding of the site's local language (e.g. Dutch, German) or English language.
* Presence of any relevant severe condition or clinically relevant abnormal laboratory parameters due to which an endoscopic or laparoscopic surgical technique is contraindicated.
* Subjects who would require an intervention to the upper mediastinum or to the upper pleural cavity regions as referred in the Senhance Surgical System User Manual (UM-001-00035_CE).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients at a participating center who have had or are scheduled to have surgery using the Senhance system
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Index surgery to 30 days postoperative
  Rate of Adverse Event (Clavien >3)
Procedure-related severe adverse event | Index surgery to 30 days post-operative
  Percent of procedurally related SAE after adjudication

SECONDARY OUTCOMES:
Length of Stay | From day of index procedure to hospital discharge, up to 2 weeks
  Total duration (in days) of hospitalization related to the index surgical procedure
Conversion to unplanned open surgery | Intraoperative (during index surgical procedure)
  Rate of unplanned conversions from laparoscopic to open surgery.
COMFORT-B scale for assessing pain in pediatric patients aged 0 to less than 2 years of age | Day after index surgery to day of discharge from hospital for index surgery, up to 2 weeks.
  The COMFORT-B Score is a validated behavioral assessment tool designed to evaluate the level of sedation, pain, and distress in pediatric patients. The COMFORT-B scale will be used to assess pain levels in children aged 0 to less than 2 years of age. The COMFORT-B scale includes six behavioral dimensions: Alertness, Calmness/Agitation, Respiratory Response (only in mechanically ventilated children), Crying (only in spontaneously breathing children), Physical Movement, Muscle Tone, and Facial Tension. Each dimension is scored on a scale from 1 to 5, yielding a total score range of 6 to 30. Higher scores indicate greater distress or discomfort.
Face, Legs, Activity, Cry, Consolability (FLACC) behavioral pain scale for children aged 2 years to less than 7 years of age. | Day after index surgery to day of discharge from hospital for index surgery, up to 2 weeks.
  The FLACC scale assesses pain by observing five categories of behaviors and assigning a score of 0-2 to each category, resulting in a total score of 0-10, where a score of 10 indicates a higher level of pain.
  The following five behavioral categories are assessed: Facial expression, leg movement, Activity level, Crying, and Consolability.
  The FLACC scale will be utilized to assess pain in children aged 2 to less than 7 years of age.
Numerical Rating Scale (NRS) for assessing pain in patients aged 7 years to less than 18 years of age. | Day after index surgery to day of discharge from hospital for index surgery, up to 2 weeks.
  Pain will be assessed using a numerical rating scale (NRS) from 0 (no pain) to 10 (worst pain). The NRS scale will be used for patients aged 7 years to less than 18 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gödeke, Dr. med., Principal Investigator — Dr. von Hauner Children's Hospital
Locations (1):
- Dr. von Hauner Children's Hospital Clinic of the University of Munich, München, Germany